CLINICAL TRIAL: NCT01880372
Title: Pilot Study: The Use of Alpha Lipoic Acid for the Treatment and Prevention of Diabetic Retinopathy
Brief Title: The Use of Alpha Lipoic Acid for the Treatment and Prevention of Diabetic Retinopathy
Acronym: ALA-TPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low number of patients enrolled
Sponsor: Ferris State University (Other)
Collaborators: Retina Specialists of Michigan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FSU130106
Record Dates: First submitted 2013-06-13; First posted 2013-06-19 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Moderate Non-proliferative Diabetic Retinopathy
Keywords: Diabetes; Diabetic Retinopathy; Retinopathy; Free radical; Retinal diseases; Antioxidants; Protective agents; Thioctic acid
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy; Retinal Diseases | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alpha Lipoic Acid Assignment Group (Experimental): Alpha lipoic acid assignment group will follow routine care and receive 600 mg oral administration of lipoic acid daily.
  Interventions: Dietary Supplement: Alpha Lipoic Acid
- Alpha Lipoic Acid Control Group (No Intervention): The control group will follow routine care alone.

INTERVENTIONS:
Dietary Supplement: Alpha Lipoic Acid — Same as Arm description
  Other Names: ALA
  Arms: Alpha Lipoic Acid Assignment Group

SUMMARY:
The purpose of this study is to evaluate the role of alpha lipoic acid in patients who have moderate non-proliferative diabetic retinopathy.

The primary aim of this study is to test the hypothesis that the addition of alpha lipoic acid in a diabetic patient's therapeutic regimen can decrease the progression of diabetic retinopathy and preserve visual acuity.

DETAILED DESCRIPTION:
Increased production of free radicals and depletion of antioxidants are commonly observed in diabetic patients. Based on animal studies, increased production of free radicals tends to persist even after blood glucose is tightly controlled. The rationale of using a potent antioxidant is based on the observation that increased oxidative stress associated with hyperglycemia can contribute to cellular injury leading to apoptosis; consequently, leading to diabetic retinopathy. Evidence from animal model showed that alpha lipoic acid (a potent antioxidant) was effective for decreasing the progression of diabetic retinopathy and in reducing free radicals.

Therefore, we hypothesize that therapy that can exert a powerful antioxidant activity can provide a therapeutic modality needed to target the pathogenesis of diabetic retinopathy.

This study will be a 12-month pilot study demonstrating the role of alpha lipoic acid in patients who have moderate non-proliferative diabetic retinopathy.

Eligible patients will be randomized to two groups, treatment and control groups. Patients in the treatment group will receive 600 mg of alpha lipoic acid daily with routine care while patient in control group will only follow routine care. Optical coherence tomography (OCT)and electronic visual acuity testing algorithm (ETDRS) will be used to measure changes in retinal thickness and visual acuity respectively. Blood changes in macrophage colony stimulating factor (M-CSF), vascular endothelia growth factor (VEGF), Interferon 2 alpha, interleukin 6 and 8 will also be evaluated and compared between the two groups. Descriptive statistics and intention to treat analysis will be used to compare treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Individual with diabetes mellitus type I or type II mild to moderate non-proliferative diabetic retinopathy which will be based on ETDRS grading scale
* Patient must be 18 years and older

Exclusion Criteria:

* Patients with severe non-proliferative or proliferative diabetic retinopathy
* Patients with macular edema
* Eye diseases that may interfere with visualization of the fundus such as preretinal hemorrhage, cataract, vitreous hemorrhage
* Patient that has undergone any type of interventional therapy for diabetic retinopathy (Such as laser photocoagulation, vitrectomy)
* Amblyopia
* Glaucoma
* Patient with cataract surgery within a period of 4 months
* Patients with other retinal diseases
* Patients on chronic administration of alpha lipoic acid
* Known intolerance/hypersensitivity to alpha lipoic acid
* Patient with history of dialysis in cases of renal insufficiency and history of kidney transplantation
* Malignancies or life threatening diseases as determined by the investigators
* Current history of drug or alcohol abuse
* Pregnant and breast feeding women
* Cognitively impaired patients
* Participation in a clinical trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Decreased progression of diabetic retinopathy. | Visual examination and serum analysis will be done at baseline, 6 and 12 month
  Decreased progression of diabetic retinopathy as measured and graded by using Standard ETDRS 7 -field color stereoscopic funds photograph, and also by measuring the serum levels of interleukin 6 and 8, VEGF, interferon 2 alpha and M-CSF using ELISA technique

SECONDARY OUTCOMES:
Changes in the plasma level of glutathione as measured by ELISA technique | Serum analysis done at baseline, 6 and 12 month

OTHER OUTCOMES:
Changes in retinal thickness as measured by optical coherence tomography (OCT) | Procedure done at baseline, 6 and 12 month
Changes in visual acuity as measured by electronic visual testing algorithm | Visual examination done at baseline, 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Arinze Nkemdirim Okere, PharmD, MS, Principal Investigator — Florida A & M University, College of Pharmacy and Pharmaceutical sciences
Locations (2):
- United States (2):
  - Ferris State University, Big Rapids, Michigan
  - Retina Specialists of Michigan, Grand Rapids, Michigan

REFERENCES:
- See also: Mechanism and clinical uses of alpha lipoic acid — http://www.umm.edu/altmed/articles/alpha-lipoic-000285.htm